CLINICAL TRIAL: NCT02608905
Title: The Effect of Dapagliflozin on Inflammation and Endothelial Function
Brief Title: Effect of Dapagliflozin on Inflammation and Endothelial Function
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to difficulty with enrollment of subjects
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Mandeep Bajaj, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-35985
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 5 mg daily by mouth for 2 weeks followed by 10 mg by mouth daily for 10 weeks
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo tablets by mouth daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Patients with Type 2 diabetes will be randomized to receive dapagliflozin 5 mg daily for 2 weeks followed by10 mg daily for 10 weeks by mouth or matching placebo for 12 weeks. All subjects will receive measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, monocyte inflammation, as well as ultrasound assessment of flow-mediated dilatation (FMD) of the brachial artery at baseline and after 12 weeks of drug treatment with either dapagliflozin or placebo.
  Other Names: Farxiga
  Arms: Dapagliflozin
Drug: Placebo — Patients with Type 2 diabetes will be randomized to receive dapagliflozin 5 mg daily for 2 weeks followed by10 mg daily for 10 weeks by mouth or matching placebo for 12 weeks. All subjects will receive measurements of fasting plasma glucose, Free Fatty Acids, inflammatory markers and adipocytokines, monocyte inflammation, as well as ultrasound assessment of flow-mediated dilatation (FMD) of the brachial artery at baseline and after 12 weeks of drug treatment with either dapagliflozin or placebo.
  Arms: Placebo

SUMMARY:
Sodium-glucose cotransporter 2 (SGLT-2) inhibitors reduce hyperglycemia and improve peripheral insulin sensitivity by ameliorating glucotoxicity. Insulin resistance in type 2 diabetes (T2DM) is associated with endothelial dysfunction and vascular inflammation. Thus strategies to improve insulin sensitivity and lower glucotoxicity may improve endothelial inflammation and vascular inflammation. However, the effects of these agents on vascular inflammation and endothelial function is not known in patients with type 2 diabetes although anti-inflammatory properties have been demonstrated in various animal models. In the present study the investigators will assess if dapagliflozin treatment for 12 weeks decreases monocyte inflammation and improves endothelial function in patients with type 2 diabetes on metformin monotherapy.

DETAILED DESCRIPTION:
The insulin-resistant state of type 2 diabetes mellitus (T2DM) is largely mediated by inflammatory pathways affecting skeletal muscle which is the primary site of whole body insulin resistance. Nuclear factor kappa B (NFkappaB) regulates pro-inflammatory cytokines which ultimately impair skeletal muscle insulin signaling and fatty acid oxidation; its activity reflects overall inflammatory tone in skeletal muscle. Recent human studies confirm that NFkappaB is elevated in the skeletal muscle of T2DM human subjects. Furthermore, the same inflammatory processes and signaling impairments contribute to worsening endothelial dysfunction, which is an independent predictor for future cardiovascular events in T2DM. In addition, these SGLT-2 Inhibitors reduce body weight, visceral adiposity, systolic and diastolic blood pressure, microalbuminuria, and oxidative stress. However, there are no studies examining the effects of SGLT-2 inhibitor therapy on NFkappaB and other inflammatory mediators in humans with T2DM. Moreover, no studies have examined the effect of SGLT-2 inhibitor therapy on endothelial function in this population. In the present study the investigators will assess whether dapagliflozin treatment for 12 weeks reduces monocyte inflammation and improves endothelial dysfunction in patients with type 2 diabetes on metformin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Men and women, ages 21 to 70 years. i) Women of childbearing potential must be using an acceptable method of contraception to avoid pregnancy throughout the study in such a manner that the risk of pregnancy is minimized.

   ii) Women must not be pregnant or breastfeeding.
3. Patients with Type 2 Diabetes Mellitus with the following parameters at study entry: hemoglobin A1c ranging from 7.0% to 9.0% and a fasting blood glucose less than or equal to 200 mg/dL.
4. Patients must be on a stable dose of Metformin therapy for 3 months; the dose of metformin will not change for the duration of the study.
5. Patients are allowed, but not required, to be on statins, Angiotensin Converting Enzyme (ACE) inhibitors, and angiotensin-receptor blockers at doses that have been stable for at least the last 3 months prior to enrollment in the study. Doses will not be changed for the duration of the study.
6. Patients must have a Body Mass Index between 27-35 kg/m2
7. Patients must have a stable body weight for three months prior to enrollment in the study.
8. Patients must have a Creatinine Clearance greater than 60 mL/min (calculated by Cockcroft-Gault formula).
9. Patients must have Hematocrit greater than or equal to 34%; Serum creatinine less than1.5 mg/dl in men and 1.4 mg/dl in women and Creatinine Clearance greater than 60 ml/min; and serum aspartate aminotransferase (AST) less than 2.5 times upper limit of normal, serum alanine transaminase (ALT) less than 2.5 times upper limit of normal, serum alkaline phosphatase less than 2.5 times upper limit of normal.

Exclusion Criteria:

1. History of Type 1 diabetes mellitus
2. Women who are pregnant or breastfeeding
3. Patients receiving lipid-lowering medications other than statins within the last 3 months.
4. Patient receiving SGLT-2 inhibitors, incretin therapy, dipeptidyl peptidase 4 (DPP-4) inhibitors, thiazolidinediones, insulin, sulfonylureas, alpha-glucosidase inhibitors, corticosteroids, immunosuppressive therapy, thiazide or loop diuretics, or hormone replacement therapy within the last 3 months .
5. Patient must stop treatment with nonsteroidal anti-inflammatory drugs (NSAID) and antioxidant vitamin supplements at least one week prior to the start of the study
6. Patients with diabetic gastroparesis.
7. Patients with current tobacco use.
8. Patients with active malignancy.
9. Patients with history of urinary bladder cancer
10. Patients with a history of clinically significant heart disease, peripheral vascular disease, or pulmonary disease will not be studied
11. Subjects with a history of any serious hypersensitivity reaction to dapagliflozin.
12. Prisoners, or subjects who are involuntarily incarcerated.
13. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.
14. Patients with significant cardiac,hepatic or renal disease (Creatinine Clearance less than 60 mL/min calculated by Cockcroft-Gault formula) will be excluded.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Bajaj, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 7 | 10
Completed | 5 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 9 | 15
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 6 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Monocyte Inflammatory Protein Nuclear Factor Kappa-B (NFkappaB) (%)
Description: The percentage change in monocyte inflammatory proteins NFkappaB (%) from baseline in patients with type 2 diabetes.
Time Frame: 12 weeks
Population: The data was not collected.
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Arterial Flow Mediated Dilatation (%)
Description: The percentage change in arterial flow mediated dilation (%) from baseline as measured by ultrasound in patients with type 2 diabetes.
Time Frame: 12 weeks
Population: The data was not collected
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/7 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02608905/Prot_SAP_000.pdf